CLINICAL TRIAL: NCT07146776
Title: Evaluation of the Effect of Injectable Platelet-Rich Fibrin in the Treatment of Periodontal Intrabony Defects With Xenogenic Grafts: a Randomized Controlled Clinical Trial
Brief Title: Treatment of Intrabony Defects With Injectable Platelet-Rich Fibrin and Xenogenic Grafts
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Tuğçe Paksoy, Associate Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-19
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Periodontitis; Intrabony Periodontal Defect; Periodontal Diseases; Periodontal Defect; Periodontal Bone Loss
Keywords: i-prf; injectable prf; injectable platelet rich fibrin; xenogenic graft; xenogenic bone graft; xenograft
MeSH Terms: conditions — Periodontitis; Periodontal Diseases; Alveolar Bone Loss | interventions — proliferation regulatory factors, human urine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- i-PRF and xenogenic graft (Experimental): In this treatment protocol, bone graft and i-PRF will be used instead of physiological saline. The preparation time for i-PRF (centrifugation) is 3 minutes. Two 9-mL tubes of venous blood will be collected from each patient.
  Interventions: Procedure: open flap debridement with I-prf and xenogeneic graft
- Saline and xenogenic graft (Active Comparator): A bovine-derived xenogeneic bone graft, which is routinely used for the treatment of intraosseous defects, will be applied. The graft will be mixed with physiological saline prior to application.
  Interventions: Procedure: open flap debridement with saline and xenogenic graft

INTERVENTIONS:
Procedure: open flap debridement with I-prf and xenogeneic graft — During the surgical phase of treatment, patients will undergo open flap debridement surgery. Infiltrative local anesthesia will first be administered to the involved teeth. The gingiva will be incised within the gingival sulcus using a scalpel, and a full-thickness flap will be carefully elevated with a periosteal elevator. Granulation tissue and dental calculus will be completely removed using Gracey curettes (American Eagle, USA) and an ultrasonic scaler. Subsequently, a xenogeneic bone graft mixed with injectable platelet-rich fibrin (i-PRF) will be applied. The flap will then be sutured using 4-0 polypropylene sutures.
  Arms: i-PRF and xenogenic graft
Procedure: open flap debridement with saline and xenogenic graft — During the surgical phase of treatment, patients will undergo open flap debridement surgery. Infiltrative local anesthesia will first be administered to the involved teeth. The gingiva will be incised within the gingival sulcus using a scalpel, and a full-thickness flap will be carefully elevated with a periosteal elevator. Granulation tissue and dental calculus will be thoroughly removed using Gracey curettes (American Eagle, USA) and an ultrasonic scaler. A xenogeneic bone graft mixed with physiological saline will then be applied. Finally, the flap will be sutured using 4-0 polypropylene sutures.
  Arms: Saline and xenogenic graft

SUMMARY:
The use of injectable platelet-rich fibrin (i-PRF) in both surgical and non-surgical dental treatments has become increasingly widespread. Hard tissue grafts can produce "sticky bone," and bone gain can have a positive effect on intrabony defects frequently seen in periodontal disease, compared to grafts alone. This study aims to clinically and radiographically evaluate the effectiveness of using bovine-derived xenogenic bone grafts in combination with i-PRF and bovine-derived xenogeneic bone grafts alone in patients with intrabony defects and stage III periodontitis.

DETAILED DESCRIPTION:
Intrabony defects are frequently observed in periodontitis patients. Bovine-derived xenogenic grafts are widely used in their treatment. To date, the graft has been mixed with various materials to increase its regenerative efficacy. In recent years, studies have explored its use in combination with PRF derivatives. Furthermore, with the introduction of i-PRF in regenerative treatments, its application with various biomaterials has been attempted. Applications have been made with materials such as demineralized freeze-dried bone allografts, hydroxyapatite bone grafts, and nanohydroxyapatite, with successful results. However, no studies have been conducted to date on the application of i-PRF with bovine-derived xenogeneic grafts in intrabony periodontal defects. This study aims to demonstrate that bovine-derived xenogeneic graft materials, which are frequently preferred by patients, achieve more successful results in various clinical and radiographic parameters in the treatment of intrabony defects, thanks to the contribution of i-PRF. The aims are to reduce clinical parameters that favor the treatment, increase bone fill, and minimize the defect area. It is thought that the use of I-PRF, a tissue-friendly biological material, will contribute to positive results in these parameters.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-65 years
* Patients with Stage III Periodontitis according to the AAP-EFP 2017 Periodontal Disease Classification
* PPD≥5 mm (if persistent 6 weeks after initial periodontal treatment)
* Intrabony defects in the interproximal region with 2 or 3 walls and a depth of at least ≥3 mm
* Non-smokers (those who smoke up to 10 per day may be included)

Exclusion Criteria:

* Patients under 18 years of age or older than 65 years of age
* Patients unable to consent
* Systemic diseases that could affect the success of surgery, such as uncontrolled diabetes
* Single-walled intrabony defects
* Those who have taken antibiotics, anti-inflammatory or immunosuppressive drugs, or birth control pills within the three months prior to the study
* Those who have received active periodontal treatment within the last six months and periodontal surgery within the last year
* Smoking more than 10 cigarettes per day
* Pregnancy or breastfeeding
* Those taking medications that affect the gums (e.g., calcium channel blockers, phenytoin or cyclosporine)
* Teeth with furcation defects
* Those undergoing active orthodontic treatment
* Those who are allergic to the biomaterials used in the study or prescribed medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-07-12 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Intrabony Defect Fill | At enrollment and 6 months control visit
  The change in the defect size will be evaluated using computed tomography. Slices with a thickness of 1.0 mm will be acquired in the sagittal plane. The defect base, alveolar bone crest, and cementoenamel junction (CEJ) will be identified on the images, and the distances between these anatomical landmarks will be measured in millimeters. The distance between the defect base and the alveolar bone crest will be used to determine the depth of the intraosseous defect.
Clinical Attachment Level | At enrollment, 3 and 6 months control visits
  It represents the value obtained by measuring the distance between the pocket base and the cementoenamel junction (CEJ) using a standard periodontal probe with a diameter of 0.4-0.5 mm, rounded to the nearest millimeter. The changes in clinical attachment level will be measured at baseline, as well as at the 3- and 6-month follow-up visits.

SECONDARY OUTCOMES:
Probing Pocket Depth | At enrollment, 3 and 6 months control visits
  Probing pocket depth, defined as the distance between the base of the periodontal pocket and the free gingival margin, is one of the important clinical parameters used to monitor tissue healing after periodontal treatments. It will be measured in mm from the six surfaces of the involved tooth (buccal mesial, buccal middle, buccal distal, palatal/lingual mesial, palatal/lingual middle, and palatal/lingual distal) using a Williams or UNC-15 periodontal probe. Changes in probing pocket depth will be recorded at baseline, as well as at the 3- and 6-month follow-up visits.
Plaque Index | At enrollment, 3 and 6 months control visits
  Patients' plaque indices will be recorded according to the Silness & Löe Index. After the teeth are air-dried, the amount of plaque near the gingival margin of each tooth will be examined with an inspection and a periodontal probe. Index values ranging from 0 to 3 are assigned based on the amount of plaque on the tooth surface. Based on this index:
  0: No plaque
  1. A thin layer of plaque is observed along the gingival margin. This thin layer can be detected with a periodontal probe.
  2. A moderate layer of plaque is observed along the gingival margin. This plaque can be visually detected.
  3. A considerable layer of plaque is observed at the gingival margin. The interdental spaces appear to be full of plaque.
Gingival Index | At enrollment, 3 and 6 months control visits
  This index was developed by Löe & Silness. This system evaluates bleeding, the most fundamental sign of inflammation. The mesial, distal, vestibular, and lingual gingiva of the teeth are evaluated. They are scored from 0 to 3. These values are then summed and divided by four. This calculates the gingival index. Dividing the total by the number of teeth yields the individual score. According to this index:
  0: Healthy gingiva, no inflammation.
  1. Mild gingival inflammation, discoloration, and mild edema. No bleeding on probing.
  2. Moderate gingival inflammation, redness, and edema. Bleeding on probing.
  3. Severe gingival inflammation, redness, and edema. Spontaneous bleeding occurs.
Pain Assasment | 2 weeks after the surgical intervention
  The Visual Analog Scale (VAS) is the most commonly used scale for both measuring pain intensity and monitoring the degree of pain relief. The VAS consists of a 10-cm line with endpoints of "no pain" and "worst possible pain." The patient marks the line that best describes their pain intensity. The average of the obtained values is calculated for each patient. The patient's pain, inability to chew, and procedural stress will be assessed with the VAS at two weeks postoperatively.
The Amount of Painkiller Used | 2 weeks after the surgical intervention
  The amount of painkiller taken after the operation will be recorded in milligram.

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bilimleri Üniversitesi, Istanbul, Üsküdar, Turkey (Türkiye)